CLINICAL TRIAL: NCT00974311
Title: Affirm: A Multinational Phase 3, Randomized, Double-blind, Placebo-controlled Efficacy And Safety Study Of Oral Mdv3100 In Patients With Progressive Castration-resistant Prostate Cancer Previously Treated With Docetaxel Based Chemotherapy
Brief Title: Safety and Efficacy Study of MDV3100 in Patients With Castration-Resistant Prostate Cancer Who Have Been Previously Treated With Docetaxel-based Chemotherapy
Acronym: AFFIRM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry); Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRPC2; 2009-013174-41 (EudraCT Number); C3431010 (Other: Alias Study Number)
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Results first posted 2012-10-30 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Castration-Resistant Prostate Cancer
Keywords: Prostate Cancer; Castration-resistant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enzalutamide (Experimental): Formerly MDV3100
  Interventions: Drug: Enzalutamide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enzalutamide — MDV3100, 160 mg orally per day
  Other Names: MDV3100; Xtandi
  Arms: Enzalutamide
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
This is a phase 3 study to compare the clinical benefit of MDV3100 versus placebo in patients with castration-resistant prostate cancer who have been previously treated with docetaxel-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Progressive prostate cancer
* Medical or surgical castration with testosterone less than 50 ng/dl
* One or two prior chemotherapy regimens. At least one chemotherapy regimen must have contained docetaxel
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate bone marrow, hepatic, and renal function
* Able to swallow the study drug and comply with study requirements
* Informed consent

Exclusion Criteria:

* Metastases in the brain or active epidural disease
* Another malignancy within the previous 5 years
* Clinically significant cardiovascular disease
* Gastrointestinal disorder affecting absorption

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1199 (Actual)
Dates: Start 2009-09-30 (Actual); Primary Completion 2011-09-15 (Actual); Study Completion 2017-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (239):
- United States (91):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Tower Cancer Research Foundation, Tower Hematology Oncology Medical Group, Beverly Hills, California
  - USC Westside Prostate Cancer Center, Beverly Hills, California
  - City of Hope, Duarte, California
  - Cancer Center Oncology Medical Group, La Mesa, California
  - LAC & USC Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - c/o Prostate Oncology Specialist, Inc., Marina del Rey, California
  - North County Oncology Medical Clinic, Inc,, Oceanside, California
  - Medical Oncology Associates - SD, San Diego, California
  - Sharp Memorial Hospital Investigational Pharmacy, San Diego, California
  - Sharp Rees-Stealy, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - City of Hope Medical Group, South Pasadena, California
  - Stanford Hospital and Clinics Research Pharmacy, Stanford, California
  - Stanford University Medical Center, Stanford, California
  - Research Pharmacist, Aurora, Colorado
  - University of Colorado Denver, Anschutz Cancer Pavilion, Aurora, Colorado
  - C/O: Thomas Ferencz R.Ph., BCOP, New Haven, Connecticut
  - Yale University School of Med, New Haven, Connecticut
  - George Washington University-Medical Faculty Associates, Washington D.C., District of Columbia
  - Palm Beach Cancer Institute, Atlantis, Florida
  - Palm Beach Cancer Institute, Palm Beach Gardens, Florida
  - Palm Beach Cancer Institute, Wellington, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Peachtree Hematology-Oncology Consultants, P.C., Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Brigham & Women's Hospital (BWH), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Siteman Cancer Center, City of Saint Peters, Missouri
  - Siteman Cancer Center-West County, Creve Coeur, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Institute, an affiliate of the UC San Diego Health System, Las Vegas, Nevada
  - New Mexico Oncology Hematology Consultants, Ltd., Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Pharmaceutical Research Services, Durham, North Carolina
  - Portland VA Medical Center, Portland, Oregon
  - UPMC Cancer Centers, McKeesport, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Hollings Cancer Center, Charleston, South Carolina
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Grand Strand Urology, Myrtle Beach, South Carolina
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Dickson, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
  - Parkland Health and Hospital System, Dallas, Texas
  - Texas Oncology, Sammons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Virginia Oncology Associates, Chesapeake, Virginia
  - Virginia Oncology Associates, Hampton, Virginia
  - Virginia Cancer Institute, Mechanicsville, Virginia
  - Virginia Cancer Institute, Midlothian, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - Virginia Oncology Associates, Williamsburg, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Argentina (10):
  - Instituto Medico de Asistencia e Investigaciones S.A (IMAI Research), Buenos Aires, AR
  - Instituto Oulton, Córdoba, Córdoba Province
  - Clinica Universitaria Privada Reina Fabiola, Córdoba, Córdoba Province
  - Policlinico Neuquen, Neuquén, Neuquén Province
  - Policlinico Modelo de Cipolletti, Cipolletti, Río Negro Province
  - Instituto de Investigaciones Clinicas Cipolletti, Cipolletti, Río Negro Province
  - Sanatorio Mapaci, Rosario, Santa Fe Province
  - Instituto de Oncologia y Especialidades Medicas, Rosario, Santa Fe Province
  - Hospital Italiano Garibaldi, Rosario, Santa Fe Province
  - Centro de Diagnostico Dr. Enrique Rossi, Buenos Aires
- Australia (29):
  - North Coast Cancer Institute, Coffs Harbour, New South Wales
  - Sydney Cancer Centre, Concord, New South Wales
  - Mid North Coast Diagnostic Imaging, Port Macquarie, New South Wales
  - Port Macquarie Base Hospital Pharmacy, Port Macquarie, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Prince of Wales Hospital, Department of Medical Oncology, Randwick, New South Wales
  - The Tweed Hospital, Tweed Heads, New South Wales
  - PRP Diagnostic Imaging, Wentworthville, New South Wales
  - Sydney West Cancer Trials Centre, Department of Medical Oncology, Westmead, New South Wales
  - River City Pharmacy, Auchenflower, Queensland
  - Heart Care Partners, Auchenflower, Queensland
  - Icon Cancer Care Wesley, Auchenflower, Queensland
  - Icon Cancer Care Chermside, Chermside, Queensland
  - Southern X-Ray Chermside, Chermside, Queensland
  - Cancer Care Services, Herston, Queensland
  - Icon Cancer Foundation, Milton, Queensland
  - Icon Cancer Care South Brisbane, South Brisbane, Queensland
  - Mater Private Cardiology, South Brisbane, Queensland
  - Queensland X-Ray, South Brisbane, Queensland
  - XRadiology, Toowong, Queensland
  - Department of Medical Oncology, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Peninsula Oncology Centre, Frankston, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Sir Charles Gairdner Hospital, Department of Medical Oncology, Nedlands, Western Australia
  - 60 Eleanor St, Footscray
  - Western Hospital, Footscray
  - The Royal Melbourne Hospital, Victoria
- Austria (3):
  - Krankenhaus der Barmherzigen Schwestern Linz, Linz
  - ISOTOPIX Ambulatorium fuer, Vienna
  - Medical University of Vienna, Vienna
- Belgium (7):
  - Cliniques Universitaires Saint- Luc, Brussels
  - AZ Sint- Lucas, Ghent
  - VZW Jessa Ziekenhuis, Hasselt
  - AZ Groeninge - Campus Kennedylaan, Kortrijk
  - AZ Groeninge - Campus Sint Maarten, Kortrijk
  - University Hospital Gasthuisberg, Leuven
  - H.-Hartziekenhuis Roeselare-Menen vzw, Roeselare
- Canada (15):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Tom Baker Cancer Centre - Holy Cross Site, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Centre for the Southern Interior, Kelowna, British Columbia
  - B.C. Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Centre, Victoria, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Urology Specialists., Montreal, Quebec
  - Imagerie medicale de la Capitale, Québec, Quebec
  - CHU de Quebec, Québec, Quebec
  - Centre de rechereche clinique et evaluative en oncologie, Québec, Quebec
- Chile (4):
  - Hospital San Jose, Santiago
  - Instituto Nacional del Cancer, Santiago
  - Centro Investigacion Clinica del Sur, Temuco
  - Instituto Oncologico, Viña del Mar
- France (22):
  - Centre Paul Papin, Angers
  - Institut Bergonie, Bordeaux
  - Centre Regional Francois Baclesse de lutte contre le cancer, Caen
  - Centre hospitalier de Cannes, Cannes
  - CHU Henri Mondor, Créteil
  - Centre Hospitalier Intercommunal Frejus-Saint Raphael, Fréjus
  - Centre hospitalier departemental Vendee, La Roche-sur-Yon
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans
  - Groupement Hospitalier Edouard Herriot - Pavillon V, Lyon
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut Curie, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Centre Hospitalier Lyon sud, Pierre-Bénite
  - CHU La Miletrie, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Hospitalier, Saint-Etienne
  - Centre d'Investigation Clinique, (CIE3), Saint-Etienne
  - Centre Rene Gauducheau, Saint-Herblain
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez
  - Hopital Foch, Suresnes
  - Institut Gustave Roussy, Villejuif
- Germany (21):
  - Universitaetsklinikum Aachen, Aachen
  - Charite - Universitaetsmedizin Berlin-Campus Benjamin Franklin, Berlin
  - Gemeinschaftspraxis Fuer Nuklearmedizin, Berlin
  - Radiologische Gemeinschaftspraxis, Berlin
  - FacharztzentrumInnere Medizin, Berlin
  - Praxis Dr. Wolfgang Hoelzer, Berlin
  - Staedtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Technical University Dresden, Dresden
  - Martini-Klinik am UKE GmbH, Hamburg
  - Roentgenpraxis, Hamburg
  - Urologische Gemeinschaftspraxis Poppenbuettel, Hamburg
  - Medizinische Hochschule Hannover - Klinik fuer Urologie und Urologische Onkologie, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Mannheim, Mannheim
  - Universitaetsklinikum Muenster, Klinik fuer Klinische Radiologie, Münster
  - Universitaetsklinikum Muenster, Klinik und Poliklinik fuer Nuklearmedizin, Münster
  - Universitaetsklinikum Muenster, Klinik und Poliklinik fuer Urologie, Münster
  - Abt.f.Diagnostische u. Interventionelle Radiologie, Tübingen
  - Klinik fuer Urologie, Tübingen
  - Nuklearmedizin, Tübingen
- Italy (4):
  - Azienda Ospedaliero-Universitaria di Modena Policlinico, Via Del Pozzo 71, Modena
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano, TO
  - Azienda Ospedaliera "Istituti Ospitalieri" di Cremona, Cremona
  - Azienda Ospedaliera San Camillo Forlanini, Rome
- Netherlands (3):
  - VU Medisch Centrum, Amsterdam
  - UMC St. Radboud, Nijmegen
  - Erasmus MC, Rotterdam
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Regionalny Szpital Specjalistyczny im. Dr. Wladyslawa Bieganskiego, Grudziądz
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika, Regionalny Osrodek Onkologiczny, Lodz
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika, Lodz
  - Wojewodzki szpital specjalistyczny im. Janusza Korczaka, Słupsk
- South Africa (3):
  - Hopelands Cancer Centre, Durban
  - GVI Oncology, Port Elizabeth
  - Sandton Oncology Centre, Sandton
- Spain (7):
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Radiodiagnostic Cetir Clinica Pilar, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Madrid Norte Sanchinarro, Madrid
  - Clinica Universidad de Navarra, Pamplona
- United Kingdom (15):
  - Bishops Wood Hospital, Northwood, Middlesex
  - Mount Vernon Hospital, Northwood, Middlesex
  - The Royal Marsden Hospital, Sutton, Surrey
  - Belfast City Hospital, Belfast
  - Cancer Centre, Birmingham
  - Bristol Haematology & Oncology Centre, Bristol
  - Bristol Royal Infirmary, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - University College Hospital, London
  - Hammersmith Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Northern Centre for Cancer Care, Newcastle upon Tyne
  - Churchill Hospital, Oxford
  - The Manor Hospital Oxford, Oxford

REFERENCES:
- [Derived] Cella D, Ganguli A, Turnbull J, Rohay J, Morlock R. US Population Reference Values for Health-Related Quality of Life Questionnaires Based on Demographics of Patients with Prostate Cancer. Adv Ther. 2022 Aug;39(8):3696-3710. doi: 10.1007/s12325-022-02204-3. Epub 2022 Jun 22. PMID 35731340
- [Derived] Joshua AM, Armstrong A, Crumbaker M, Scher HI, de Bono J, Tombal B, Hussain M, Sternberg CN, Gillessen S, Carles J, Fizazi K, Lin P, Duggan W, Sugg J, Russell D, Beer TM. Statin and metformin use and outcomes in patients with castration-resistant prostate cancer treated with enzalutamide: A meta-analysis of AFFIRM, PREVAIL and PROSPER. Eur J Cancer. 2022 Jul;170:285-295. doi: 10.1016/j.ejca.2022.04.005. Epub 2022 May 26. PMID 35643841
- [Derived] Zhao JL, Fizazi K, Saad F, Chi KN, Taplin ME, Sternberg CN, Armstrong AJ, de Bono JS, Duggan WT, Scher HI. The Effect of Corticosteroids on Prostate Cancer Outcome Following Treatment with Enzalutamide: A Multivariate Analysis of the Phase III AFFIRM Trial. Clin Cancer Res. 2022 Mar 1;28(5):860-869. doi: 10.1158/1078-0432.CCR-21-1090. PMID 34965947
- [Derived] Tombal BF, Freedland SJ, Armstrong AJ, Beer TM, Stenzl A, Sternberg CN, Hussain M, Ganguli A, Ramaswamy K, Bhadauria H, Ivanescu C, Turnbull J, Holmstrom S, Saad F. Impact of enzalutamide on patient-reported fatigue in patients with prostate cancer: data from the pivotal clinical trials. Prostate Cancer Prostatic Dis. 2022 Feb;25(2):288-295. doi: 10.1038/s41391-021-00447-9. Epub 2021 Sep 13. PMID 34518652
- [Derived] Armstrong AJ, Al-Adhami M, Lin P, Parli T, Sugg J, Steinberg J, Tombal B, Sternberg CN, de Bono J, Scher HI, Beer TM. Association Between New Unconfirmed Bone Lesions and Outcomes in Men With Metastatic Castration-Resistant Prostate Cancer Treated With Enzalutamide: Secondary Analysis of the PREVAIL and AFFIRM Randomized Clinical Trials. JAMA Oncol. 2020 Feb 1;6(2):217-225. doi: 10.1001/jamaoncol.2019.4636. PMID 31830211
- [Derived] Poon DMC, Wong KCW, Chan TW, Law K, Chan K, Lee EKC, Lee C, Chan M; Hong Kong Society of Uro-Oncology (HKSUO). Survival Outcomes, Prostate-specific Antigen Response, and Tolerance in First and Later Lines of Enzalutamide Treatment for Metastatic Castration-resistant Prostate Cancer: A Real-World Experience in Hong Kong. Clin Genitourin Cancer. 2018 Oct;16(5):402-412.e1. doi: 10.1016/j.clgc.2018.07.008. Epub 2018 Jul 21. PMID 30126765
- [Derived] Heller G, McCormack R, Kheoh T, Molina A, Smith MR, Dreicer R, Saad F, de Wit R, Aftab DT, Hirmand M, Limon A, Fizazi K, Fleisher M, de Bono JS, Scher HI. Circulating Tumor Cell Number as a Response Measure of Prolonged Survival for Metastatic Castration-Resistant Prostate Cancer: A Comparison With Prostate-Specific Antigen Across Five Randomized Phase III Clinical Trials. J Clin Oncol. 2018 Feb 20;36(6):572-580. doi: 10.1200/JCO.2017.75.2998. Epub 2017 Dec 22. PMID 29272162
- [Derived] Antoun S, Bayar A, Ileana E, Laplanche A, Fizazi K, di Palma M, Escudier B, Albiges L, Massard C, Loriot Y. High subcutaneous adipose tissue predicts the prognosis in metastatic castration-resistant prostate cancer patients in post chemotherapy setting. Eur J Cancer. 2015 Nov;51(17):2570-7. doi: 10.1016/j.ejca.2015.07.042. Epub 2015 Aug 13. PMID 26278649
- [Derived] Gibbons JA, Ouatas T, Krauwinkel W, Ohtsu Y, van der Walt JS, Beddo V, de Vries M, Mordenti J. Clinical Pharmacokinetic Studies of Enzalutamide. Clin Pharmacokinet. 2015 Oct;54(10):1043-55. doi: 10.1007/s40262-015-0271-5. PMID 25917876
- [Derived] Cella D, Ivanescu C, Holmstrom S, Bui CN, Spalding J, Fizazi K. Impact of enzalutamide on quality of life in men with metastatic castration-resistant prostate cancer after chemotherapy: additional analyses from the AFFIRM randomized clinical trial. Ann Oncol. 2015 Jan;26(1):179-185. doi: 10.1093/annonc/mdu510. Epub 2014 Oct 30. PMID 25361992
- [Derived] Saad F, de Bono J, Shore N, Fizazi K, Loriot Y, Hirmand M, Franks B, Haas GP, Scher HI. Efficacy outcomes by baseline prostate-specific antigen quartile in the AFFIRM trial. Eur Urol. 2015 Feb;67(2):223-30. doi: 10.1016/j.eururo.2014.08.025. Epub 2014 Aug 27. PMID 25171902
- [Derived] Merseburger AS, Scher HI, Bellmunt J, Miller K, Mulders PF, Stenzl A, Sternberg CN, Fizazi K, Hirmand M, Franks B, Haas GP, de Bono J, de Wit R. Enzalutamide in European and North American men participating in the AFFIRM trial. BJU Int. 2015 Jan;115(1):41-9. doi: 10.1111/bju.12898. Epub 2014 Oct 23. PMID 25123978
- [Derived] Fizazi K, Scher HI, Miller K, Basch E, Sternberg CN, Cella D, Forer D, Hirmand M, de Bono JS. Effect of enzalutamide on time to first skeletal-related event, pain, and quality of life in men with castration-resistant prostate cancer: results from the randomised, phase 3 AFFIRM trial. Lancet Oncol. 2014 Sep;15(10):1147-56. doi: 10.1016/S1470-2045(14)70303-1. Epub 2014 Aug 4. PMID 25104109
- [Derived] Scher HI, Fizazi K, Saad F, Taplin ME, Sternberg CN, Miller K, de Wit R, Mulders P, Chi KN, Shore ND, Armstrong AJ, Flaig TW, Flechon A, Mainwaring P, Fleming M, Hainsworth JD, Hirmand M, Selby B, Seely L, de Bono JS; AFFIRM Investigators. Increased survival with enzalutamide in prostate cancer after chemotherapy. N Engl J Med. 2012 Sep 27;367(13):1187-97. doi: 10.1056/NEJMoa1207506. Epub 2012 Aug 15. PMID 22894553

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1199 participants were enrolled and randomized for double-blind (DB) phase. Out of which, 159 participants entered the optional open-label extension (OLE) phase.
Pre-assignment Details: Participants were randomized 2:1 to receive either Enzalutamide or Placebo in DB phase. All participants who continued in OLE phase, received Enzalutamide.
Groups:
- Enzalutamide: In DB Phase, participants received Enzalutamide capsules 160 mg orally per day. Participants who completed DB Phase, entered in optional OLE Phase and received same treatment until unacceptable toxicity, confirmed disease progression and the participant was scheduled to initiate a new systemic anti-neoplastic therapy, death or withdrawal (median treatment duration was 8.3 months).
- Placebo: In DB Phase, participants received placebo capsules (for Enzalutamide) orally per day. Participants who completed DB Phase, entered in optional OLE Phase and received Enzalutamide capsules 160 mg orally per day until unacceptable toxicity, confirmed disease progression and the participant was scheduled to initiate a new systemic anti-neoplastic therapy, death or withdrawal (median treatment duration was 3.0 months in DB Phase and 7.7 months in OLE Phase).
Period: DB Phase (up to 24 Months)
Arm/Group | Enzalutamide | Placebo
Started | 800 | 399
Completed | 109 | 50
Not Completed | 691 | 349
Not completed — Lost to Follow-up | 5 | 2
Not completed — Death | 561 | 298
Not completed — Withdrawal by Subject | 16 | 7
Not completed — Study Terminated by Sponsor | 108 | 42
Not completed — Other | 1 | 0
Period: OLE Phase (up to 77 Months)
Arm/Group | Enzalutamide | Placebo
Started | 109 | 50
Completed | 0 | 0
Not Completed | 109 | 50
Not completed — Death | 14 | 21
Not completed — Study Terminated by Sponsor | 78 | 26
Not completed — Other | 15 | 2
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population (ITT) included all participants who were randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Enzalutamide | Placebo | Total
Number analyzed (Participants) | 800 | 399 | 1199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 232 | 130 | 362
  >=65 years | 568 | 269 | 837
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (7.96) | 68.6 (8.39) | 68.7 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 800 | 399 | 1199
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 23 | 55
  Not Hispanic or Latino | 768 | 376 | 1144
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 5 | 8 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 27 | 20 | 47
  White | 745 | 366 | 1111
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 21 | 4 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 181 | 107 | 288
  Spain | 23 | 13 | 36
  Austria | 15 | 10 | 25
  Chile | 6 | 5 | 11
  United Kingdom | 82 | 50 | 132
  Italy | 20 | 10 | 30
  France | 193 | 80 | 273
  Canada | 82 | 25 | 107
  Argentina | 7 | 3 | 10
  Belgium | 27 | 18 | 45
  Poland | 7 | 4 | 11
  Australia | 60 | 33 | 93
  South Africa | 3 | 3 | 6
  Germany | 62 | 24 | 86
  Netherlands | 32 | 14 | 46

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Survival was defined as time from randomization to death due to any cause. The duration of overall survival was right-censored for participants who were lost to follow-up since randomization or not known to have died at the data analysis cut-off date (this included participants who were known to have died after the data analysis cut-off date).
Time Frame: During study period (up to 101 months)
Population: ITT included all participants who were randomized into the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 800 | 399
Months | 18.4 [17.3 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment | 13.6 [11.3 to 15.8]
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank; Stratified by baseline Eastern Cooperative Oncology Group (ECOG) performance status and mean Brief Pain Inventory - Short Form score (Question #3); Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.53 to 0.75] — Hazard Ratio and 95% confidence interval are from Cox regression model

2. Secondary Outcome: Radiographic Progression-free Survival
Description: Radiographic progression-free survival was defined as time from randomization to the earliest objective evidence of radiographic progression or death due to any cause. Participants were assessed for objective disease progression at regularly scheduled visits. The consensus guidelines of the Prostate Cancer Clinical Trials Working Group 2 were taken into consideration for the determination of disease progression. Radiographic disease progression was defined by Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 for soft tissue disease, or the appearance of two or more new bone lesions on bone scan. Progression at the first scheduled reassessment at Week 13 required a confirmatory scan 6 or more weeks later. Participants who did not reach the endpoint were right censored at their last assessment.
Time Frame: During DB phase (up to 24 months)
Population: ITT included all participants who were randomized into the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 800 | 399
Months | 8.3 [8.2 to 9.4] | 2.9 [2.8 to 3.4]
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank; Stratified by baseline ECOG performance status and mean Brief Pain Inventory - Short Form score (Question #3); Hazard Ratio (HR) = 0.40, 95% CI 2-sided [0.35 to 0.47] — Hazard Ratio and 95% confidence interval are from Cox regression model

3. Secondary Outcome: Time to First Skeletal-related Event
Description: The time to first skeletal-related event was defined as time from randomization to the occurrence of the first skeletal-related event. Participants were assessed for skeletal-related events at regularly scheduled visits. A skeletal-related event was defined as radiation therapy or surgery to bone, pathologic bone fracture, spinal cord compression, or change of antineoplastic therapy to treat bone pain. Participants who did not reach the endpoint were right censored at their last assessment.
Time Frame: During DB Phase (up to 24 months)
Population: ITT included all participants who were randomized into the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 800 | 399
Months | 16.7 [14.6 to 19.1] | 13.3 [9.9 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority or Other; p = 0.0001, Log Rank; Stratified by baseline ECOG performance status and mean Brief Pain Inventory - Short Form score (Question #3); Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.566 to 0.835] — Hazard Ratio and 95% confidence interval are from Cox regression model

4. Secondary Outcome: Percentage of Participants Who Were Responders for Functional Assessment of Cancer Therapy-Prostate (FACT-P)
Description: The FACT-P was a 39-item participant questionnaire which assessed physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and additional prostate cancer specific concerns (12 items). All items were scored from 0 (not at all) to 4 (very much). The sum of scores on all 5 domains constitutes the global FACT-P. The global/total FACT-P score ranged from 0 (worst) to 156 (best), higher scores indicate better health status. Responders were those participants who had a 10-point improvement in their total FACT-P score, as compared with baseline, on two consecutive measurements obtained at least 3 weeks apart.
Time Frame: Baseline up to 24 months
Population: Evaluable intent to treat (ITT) - all participants who were part of the ITT population and had a global FACT-P score at baseline and at least 1 post-baseline assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 651 | 257
Percentage of participants | 43.2 [39.3 to 47.1] | 18.3 [13.8 to 23.6]
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by baseline ECOG performance status and mean Brief Pain Inventory - Short Form score (Question #3); Difference in Percentage of Participants = 24.9, 95% CI 2-sided [18.8 to 30.9] — Confidence Interval based on standard normal approximation

5. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: Time to PSA progression was defined as time from randomization to PSA progression. Participants who did not reach the endpoint were right censored at their last assessment or for participants with no post-baseline PSA assessment, date of randomization. For participants with PSA declines at Week 13, the PSA progression date was defined as the date that a >=25% increase and an absolute increase of >=2 nanogram per milliliter (ng/mL) above the nadir was documented, which was confirmed by a second consecutive value obtained 3 or more weeks later (required only if PSA progression did not occur at last PSA assessment). For participants with no PSA declines at Week 13, PSA progression date was defined as the date that a >=25% increase and an absolute increase of >=2 ng/mL above the baseline was documented, which was confirmed by a second consecutive value 3 or more weeks later (required only if PSA progression did not occur at last PSA assessment).
Time Frame: Baseline and at every study visit from Week 13 while on study drug (up to 24 months)
Population: ITT included all participants who were randomized into the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 800 | 399
Months | 8.3 [5.8 to 8.3] | 3.0 [2.9 to 3.7]
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — Stratified by baseline ECOG performance status and mean Brief Pain Inventory - Short Form score (Question #3); Hazard Ratio (HR) = 0.248, 95% CI 2-sided [0.204 to 0.303] — Hazard Ratio and 95% confidence interval are from Cox regression model

6. Secondary Outcome: Percentage of Participants With Pain Palliation
Description: The proportion of participants with pain palliation was assessed for participants with a stable and sufficient pain burden at study entry. Pain burden was measured by question #3 of the Brief Pain Inventory (Short Form). This scale measures pain on a 0 to 10 scale with 0 indicating no pain and 10 indicating pain as bad as you can imagine. Pain palliation at Week 13 was determined for the proportion of men with baseline bone metastasis(es) who had baseline pain attributable to the metastasis(es). Palliation was defined as >=30% reduction in average pain score at Week 13 compared to baseline without a >=30% increase in analgesic use.
Time Frame: Baseline up to 24 months
Population: Evaluable ITT Population included participants with metastatic bone disease at baseline; provided answers to Question #3 of the Brief Pain Inventory - Short Form for a minimum of 4 out of 7 days in the baseline run-in period; stable baseline pain; stable analgesic use; and had an average pain score during the baseline run-in period of >= 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 49 | 15
Percentage of participants | 44.9 [30.7 to 59.8] | 6.7 [0.2 to 31.9]
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority or Other; p = 0.0079, Cochran-Mantel-Haenszel; Stratified by baseline Eastern Cooperative Oncology Group performance status (0-1 vs. 2); Difference in Rate of Pain Palliation = 38.2, 95% CI 2-sided [19.4 to 57.0] — Confidence Interval based on standard normal approximation

7. Secondary Outcome: Percentage of Participants With Prostate Specific Antigen (PSA) Response
Description: Participants were evaluable for PSA response rate if they had a PSA level measured at baseline and at least 1 post-baseline assessment. Both PSA responses of > 50% and > 90% were determined. PSA responses required confirmation with a subsequent assessment that was conducted at least 3 weeks later.
Time Frame: During DB phase (up to 24 months)
Population: Evaluable ITT population included participants who were part of the ITT Population and had a PSA level measured at baseline and at least 1 post-baseline assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 731 | 330
Percentage of participants
  Decline >=50% from baseline | 54 | 2
  Decline >=90% from baseline | 25 | 1

8. Secondary Outcome: Percentage of Participants With Soft-tissue Objective Response
Description: The best overall soft tissue response as assessed using RECIST v1.1 during the study was summarized using the investigators' response assessments and also the derived response assessments by treatment group. Only participants with measurable soft tissue disease at screening were included in this analysis. Participants with measurable disease at screening are participants who had at least 1 target lesion identified per RECIST v1.1 at screening. Percentage of participants summarizes the number of participants with complete or partial objective response (%). Soft Tissue assessment based on Eisenhauer EA, Therasse P, Bogaerts J et al. New response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1). Eur J Cancer 2009; 45:228-247.
Time Frame: During DB phase (up to 24 months)
Population: ITT with measurable disease population included participants who were part of the ITT Population and had measurable soft tissue disease at screening, defined by at least 1 target lesion according to RECIST v1.1.
Measure: Number; unit: Percentage of participants
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 446 | 208
Percentage of participants | 29 | 4

9. Secondary Outcome: European Quality of Life Five-Domain (EQ-5D) Scale
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility or index score. Five parameters (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) were assessed on 3-point categorical scale (1= no problems, 2= some/moderate problems and 3= severe problem). Score were transformed and resulted in a total EQ-5D score range of 0 (worst imaginable health state) to 100 (best imaginable health state), with higher scores indicating better health and quality of life.
Time Frame: Week 13
Population: Evaluable ITT included participants who were part of the ITT Population and who were evaluable for EQ-5D.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 126 | 55
units on a scale | 67.2 (19.29) | 60.0 (19.26)

10. Secondary Outcome: Percentage of Participants With Circulating Tumor Cell (CTC) Conversion
Description: CTC conversion was assessed for participants with baseline CTC counts of greater than or equal to (>=) 5 cells per 7.5 milliliter (mL) of blood. A CTC conversion was defined as a decline in the CTC count to less than (<) 5 cells per 7.5 mL of blood. In this outcome measure percentage of participants with CTC conversion was reported.
Time Frame: Baseline up to 24 months
Population: CTC evaluable population included participants with a baseline and at least 1 post baseline CTC assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 127 | 62
percentage of participants | 48 [39.09 to 57.07] | 9.7 [3.63 to 19.88]

11. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE: AE resulting in any of following outcomes or deemed significant and jeopardized participants or required treatment to prevent other AE outcomes for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were events which occurred between first dose of study drug and up to the safety follow-up visit or the initiation of another anti-neoplastic therapy, whichever occurred first (up to 101 months). AEs included both serious and non-serious AEs. Clinically significant physical examination abnormalities were reported as AEs. Unscheduled visit was performed at any time during the study whenever necessary to assess for or follow-up on AEs, at the participant's request or if deemed necessary by the investigator.
Time Frame: Baseline, up to the safety follow-up visit or unscheduled visit or the initiation of another anti-neoplastic therapy whichever occurred first (up to 101 months)
Population: Safety population was defined as all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: DB Phase: In DB Phase, participants received placebo capsules (for Enzalutamide) orally per day until unacceptable toxicity, confirmed disease progression and the participant was scheduled to initiate a new systemic anti-neoplastic therapy, death or withdrawal (median treatment duration was 3.0 months).
- Placebo (DB) /Enzalutamide 160 mg (OLE) Phase: Participants who received placebo in DB phase, completed DB Phase and entered in optional OLE Phase, received Enzalutamide capsules 160 mg orally per day until unacceptable toxicity, confirmed disease progression and the participant was scheduled to initiate a new systemic anti-neoplastic therapy, death or withdrawal (median treatment duration was 7.7 months).
Arm/Group | Enzalutamide | Placebo: DB Phase | Placebo (DB) /Enzalutamide 160 mg (OLE) Phase
Number analyzed (Participants) | 800 | 399 | 50
Participants
  AEs | 789 | 390 | 48
  SAEs | 319 | 155 | 25

12. Other Pre Specified Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Criteria for abnormalities in vital signs included: sitting/supine systolic blood pressure (SBP) values: absolute result greater than (>) 180 millimeter of mercury (mmHg) and >40 mmHg increase from baseline (BL) and less than (<) 90 mmHg and >30 mmHg decrease from BL; diastolic blood pressure (DBP) values: absolute result >105 mmHg and >30 mmHg increase from BL and absolute result < 50 mmHg and >20 mmHg decrease from BL; any abnormalities in SBP or DBP; heart rate values: absolute result > 120 beats per minute (bpm) and >30 bpm increase from BL and absolute result < 50 bpm and >20 bpm decrease from BL or any abnormalities in heart rate. Unscheduled visit was performed at any time during the study whenever necessary to assess for or follow-up on AEs, at the participant's request or if deemed necessary by the investigator.
Time Frame: as for outcome 11
Population: Safety population was defined as all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide | Placebo: DB Phase | Placebo (DB) /Enzalutamide 160 mg (OLE) Phase
Number analyzed (Participants) | 800 | 399 | 50
Participants
  SBP: >180 mmHg and >40 mmHg Increase from BL | 28 | 7 | 1
  SBP: < 90 mmHg and >30 mmHg Decrease from BL | 13 | 5 | 0
  DBP: >105 mmHg and >30 mmHg Increase from BL | 5 | 2 | 0
  DBP: < 50 mmHg and >20 mmHg Decrease from BL | 13 | 3 | 1
  Any abnormalities in SBP or DBP | 52 | 16 | 2
  Heart Rate: > 120 bpm and >30 bpm Increase from BL | 7 | 5 | 0
  Heart Rate: < 50 bpm and >20 bpm Decrease from BL | 18 | 1 | 0
  Any abnormalities in Heart Rate | 25 | 6 | 0

13. Other Pre Specified Outcome: Number of Participants With Any Newly Clinically Significant Abnormal Finding in Electrocardiogram (ECG)
Description: Any new post baseline abnormality was defined as any abnormal ECG finding that appeared after baseline assessment which was not seen at the screening or baseline ECG assessment. Where, criteria of abnormality was QTcF interval > 470 millisecond (msec). Participants were counted once only for a specific abnormality. This outcome measure was planned to be analysed in double blind phase only. Unscheduled visit was performed at any time during the study whenever necessary to assess for or follow-up on AEs, at the participant's request or if deemed necessary by the investigator.
Time Frame: Baseline, up to the end of DB phase or unscheduled visit (up to 24 months)
Population: Safety population was defined as all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide | Placebo: DB Phase
Number analyzed (Participants) | 800 | 399
Participants | 28 | 13

14. Other Pre Specified Outcome: Number of Participants With Grade 3/4 Post-Baseline Laboratory Toxicity (Hematology and Chemistry)
Description: Laboratory parameters included hematological and chemistry parameters. Chemistry parameters included alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bilirubin, calcium, creatine kinase, creatinine, glucose, magnesium, phosphate, potassium and sodium. Hematology parameters included haemoglobin, leukocytes, lymphocytes, neutrophils and platelet. Test abnormalities were graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03 as Grade 3= severe and Grade 4= life-threatening or disabling. Only categories with at least 1 participant with abnormality are reported in this outcome measure. Unscheduled visit was performed at any time during the study whenever necessary to assess for or follow-up on AEs, at the participant's request or if deemed necessary by the investigator.
Time Frame: as for outcome 11
Population: Safety population was defined as all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide | Placebo: DB Phase | Placebo (DB) /Enzalutamide 160 mg (OLE) Phase
Number analyzed (Participants) | 800 | 399 | 50
Participants
  Alanine Aminotransferase:High | 2 | 2 | 1
  Albumin: Low | 7 | 3 | 0
  Alkaline Phosphatase: High | 102 | 74 | 3
  Aspartate Aminotransferase: High | 3 | 4 | 1
  Bilirubin: High | 2 | 0 | 0
  Calcium: Low | 14 | 15 | 1
  Calcium: High | 1 | 0 | 0
  Creatine Kinase: High | 4 | 2 | 0
  Creatinine: High | 0 | 2 | 0
  Glucose: High | 17 | 10 | 1
  Magnesium: Low | 0 | 1 | 0
  Magnesium: High | 1 | 1 | 0
  Phosphate: Low | 28 | 10 | 2
  Potassium: Low | 7 | 4 | 1
  Potassium: High | 2 | 3 | 0
  Sodium: Low | 19 | 13 | 0
  Sodium: High | 0 | 1 | 0
  Hemoglobin: Low | 38 | 20 | 4
  Hemoglobin: High | 1 | 0 | 0
  Leukocytes: Low | 8 | 1 | 1
  Lymphocytes: Low | 80 | 48 | 5
  Neutrophils: Low | 10 | 0 | 1
  Platelet; Low | 4 | 4 | 0

ADVERSE EVENTS:
Time Frame: Baseline, up to the safety follow-up visit or unscheduled visit or the initiation of another anti-neoplastic therapy whichever occurred first (up to 101 months)
Description: An event may be categorized as serious in one participant and non serious in another participant, or one participant may experience both serious and non serious event. All treatment emergent AEs and SAEs were collected and reported. The same event may appear as both AE and SAE. All-cause mortality data included all anticipated and unanticipated deaths due to any cause. Safety population included all randomized participants who received at least 1 dose of study drug.
Groups:
- Enzalutamide: DB + OLE Phase: In DB Phase, participants received Enzalutamide capsules 160 mg orally per day. Participants who completed DB Phase, entered in optional OLE Phase and received same treatment until unacceptable toxicity, confirmed disease progression and the participant was scheduled to initiate a new systemic anti-neoplastic therapy, death or withdrawal.
Arm/Group | Enzalutamide: DB + OLE Phase | Placebo: DB Phase | Placebo (DB) /Enzalutamide 160 mg (OLE) Phase
Serious Adverse Events (participants affected / at risk) | 319/800 | 155/399 | 25/50
Other Adverse Events (participants affected / at risk) | 784/800 | 385/399 | 47/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide: DB + OLE Phase (N=800) | Placebo: DB Phase (N=399) | Placebo (DB) /Enzalutamide 160 mg (OLE) Phase (N=50)
Anaemia (Blood and lymphatic system disorders) | 22 | 12 | 2
Anaemia of malignant disease (Blood and lymphatic system disorders) | 2 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 3 | 2 | 2
Angina pectoris (Cardiac disorders) | 2 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0
Mitral valve incompetance (Cardiac disorders) | 1 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 2 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0
Papilloedema (Eye disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 8 | 1
Nausea (Gastrointestinal disorders) | 5 | 3 | 1
Constipation (Gastrointestinal disorders) | 5 | 3 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal mass (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 22 | 8 | 3
Asthenia (General disorders) | 4 | 2 | 0
Pain (General disorders) | 5 | 1 | 0
Fatigue (General disorders) | 3 | 2 | 1
Pyrexia (General disorders) | 2 | 5 | 1
Oedema peripheral (General disorders) | 1 | 2 | 0
Malaise (General disorders) | 2 | 2 | 0
Chest pain (General disorders) | 1 | 1 | 0
Death (General disorders) | 1 | 0 | 0
Euthanasia (General disorders) | 0 | 1 | 0
General symptom (General disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 15 | 5 | 1
Urinary tract infection (Infections and infestations) | 9 | 5 | 1
Urosepsis (Infections and infestations) | 4 | 1 | 0
Sepsis (Infections and infestations) | 4 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0
Device related infection (Infections and infestations) | 3 | 0 | 0
Escherichia sepsis (Infections and infestations) | 2 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1 | 0
Chest wall abscess (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Extradural abscess (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Septic Shock (Infections and infestations) | 1 | 1 | 0
Tooth Infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Viral pericarditis (Infections and infestations) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 3 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 7 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 12 | 3 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 15 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 | 3 | 3
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 5 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 0
Metastases to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Acute monocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bone marrow tumour cell infiltration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 54 | 15 | 3
Cauda equina syndrome (Nervous system disorders) | 6 | 0 | 0
Nerve root compression (Nervous system disorders) | 1 | 4 | 0
Syncope (Nervous system disorders) | 5 | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 4 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 2 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 0
Transient ischemic attack (Nervous system disorders) | 3 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1 | 0
Convulsion (Nervous system disorders) | 4 | 0 | 2
Epiduritis (Nervous system disorders) | 2 | 0 | 0
Nerve compression (Nervous system disorders) | 1 | 1 | 0
Partial seizures (Nervous system disorders) | 2 | 0 | 0
Lethargy (Nervous system disorders) | 3 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0
Akathisia (Nervous system disorders) | 1 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 0
Cranial nerve palsies multiple (Nervous system disorders) | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Motor dysfunction (Nervous system disorders) | 0 | 1 | 0
Pachymeningitis (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0
Hypoglossal nerve paresis (Nervous system disorders) | 1 | 0 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0
Visual field defect (Nervous system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 2 | 2 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 2 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 18 | 5 | 1
Urinary retention (Renal and urinary disorders) | 7 | 8 | 0
Urinary tract obstruction (Renal and urinary disorders) | 8 | 1 | 0
Post renal failure (Renal and urinary disorders) | 3 | 3 | 0
Renal failure (Renal and urinary disorders) | 3 | 3 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 3 | 0
Bladder perforation (Renal and urinary disorders) | 1 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 2 | 0 | 0
Renal colic (Renal and urinary disorders) | 2 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Vascular purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Bladder catheter removal (Surgical and medical procedures) | 1 | 0 | 0
Limb operation (Surgical and medical procedures) | 1 | 0 | 0
Pain management (Surgical and medical procedures) | 1 | 0 | 0
Cataract operation (Surgical and medical procedures) | 0 | 1 | 0
Colon polypectomy (Surgical and medical procedures) | 1 | 0 | 0
Oesophageal dilation procedure (Surgical and medical procedures) | 1 | 0 | 0
Pleurodesis (Surgical and medical procedures) | 1 | 0 | 0
Ureteral stent insertion (Surgical and medical procedures) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 3 | 0
Haematoma (Vascular disorders) | 3 | 0 | 0
Lymphoedema (Vascular disorders) | 2 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Eyelid bleeding (Eye disorders) | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Proctocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Device dislocation (General disorders) | 1 | 0 | 0
Device occlusion (General disorders) | 0 | 1 | 0
Disease progression (General disorders) | 1 | 0 | 2
Local swelling (General disorders) | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Abscess jaw (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1
Atypical mycobacterial pneumonia (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0
Gas gangrene (Infections and infestations) | 1 | 0 | 0
Pleural infection (Infections and infestations) | 0 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Coagulation time prolonged (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Complex partial seizures (Nervous system disorders) | 1 | 0 | 0
Cranial nerve disorder (Nervous system disorders) | 2 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 1
Paraplegia (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Senile dementia (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Thalamic infarction (Nervous system disorders) | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide: DB + OLE Phase (N=800) | Placebo: DB Phase (N=399) | Placebo (DB) /Enzalutamide 160 mg (OLE) Phase (N=50)
Anaemia (Blood and lymphatic system disorders) | 123 | 70 | 11
Nausea (Gastrointestinal disorders) | 276 | 166 | 16
Constipation (Gastrointestinal disorders) | 209 | 109 | 7
Diarrhoea (Gastrointestinal disorders) | 180 | 70 | 9
Vomiting (Gastrointestinal disorders) | 141 | 84 | 8
Abdominal pain (Gastrointestinal disorders) | 47 | 21 | 2
Fatigue (General disorders) | 280 | 115 | 14
Asthenia (General disorders) | 148 | 67 | 9
Oedema peripheral (General disorders) | 121 | 46 | 4
Pyrexia (General disorders) | 59 | 23 | 4
Urinary tract infection (Infections and infestations) | 68 | 24 | 3
Weight decreased (Investigations) | 108 | 42 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 225 | 91 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 182 | 71 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 137 | 62 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 101 | 61 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 121 | 40 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 77 | 34 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 74 | 27 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 56 | 26 | 2
Headache (Nervous system disorders) | 101 | 21 | 1
Dizziness (Nervous system disorders) | 59 | 22 | 4
Paraesthesia (Nervous system disorders) | 53 | 18 | 1
Insomnia (Psychiatric disorders) | 71 | 24 | 2
Anxiety (Psychiatric disorders) | 55 | 16 | 6
Depression (Psychiatric disorders) | 51 | 19 | 4
Haematuria (Renal and urinary disorders) | 51 | 14 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 88 | 39 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 60 | 25 | 2
Hot flush (Vascular disorders) | 165 | 41 | 1
Hypertension (Vascular disorders) | 60 | 11 | 2
Abdominal pain upper (Gastrointestinal disorders) | 41 | 13 | 0
Pain (General disorders) | 27 | 12 | 3
Nasopharyngitis (Infections and infestations) | 47 | 12 | 2
Fall (Injury, poisoning and procedural complications) | 44 | 5 | 5
Decreased appetite (Metabolism and nutrition disorders) | 246 | 121 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 31 | 14 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 34 | 17 | 3
Hypoaesthesia (Nervous system disorders) | 33 | 7 | 4
Confusional state (Psychiatric disorders) | 23 | 9 | 3
Pollakiuria (Renal and urinary disorders) | 44 | 10 | 3

LIMITATIONS AND CAVEATS:
The primary objectives (overall survival) of the study had been met and all participants who had remained on study treatment have discontinued and therefore the study has been considered as completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.